CLINICAL TRIAL: NCT02503241
Title: Open Lung Strategy in Critically Ill Morbid Obese Patients Lung Imaging and Heart-lung Interaction
Brief Title: Open Lung Strategy in Critically Ill Morbid Obese Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Robert M. Kacmarek, RRT, PhD, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PRICESEOBESE
Record Dates: First submitted 2015-07-17; First posted 2015-07-20 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Obesity; Respiratory Insufficiency; Right-Sided Heart Failure; Pulmonary Atelectasis; Respiratory Mechanics
MeSH Terms: conditions — Obesity; Respiratory Insufficiency; Heart Failure; Pulmonary Atelectasis

STUDY DESIGN:
Intervention Model Description: Physiologic crossover study. There is no randomization. All participants will receive the same interventions in the same order.
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEEP_Titration_INCREMENTAL (Experimental): The investigators will compare 3 levels of PEEP (BASELINE versus PEEP INCREMENTAL versus PEEP DECREMENTAL). Baseline PEEP is based in the standard of care PEEP used in the participant units. PEEP incremental value is based in transpulmonary pressure.
  Intervention : PEEP INCREMENTAL
  Interventions: Procedure: PEEP INCREMENTAL; Procedure: PEEP DECREMENTAL
- PEEP_Titration_DECREMENTAL (Experimental): The investigators will compare 3 levels of PEEP (BASELINE versus PEEP INCREMENTAL versus PEEP DECREMENTAL). Baseline PEEP is based in the standard of care PEEP used in the participant units. PEEP decremental value is based in lung recruitment maneuver followed by a best compliance curve during PEEP decrements.
  Intervention :PEEP DECREMENTAL
  Interventions: Procedure: PEEP INCREMENTAL; Procedure: PEEP DECREMENTAL

INTERVENTIONS:
Procedure: PEEP INCREMENTAL — PEEP was progressively increased by steps of 2 cmH2O every 60 second until the end-expiratory transpulmonary pressure became positive between 0-2 cmH2O.
  Other Names: PEEP_Titration
Procedure: PEEP DECREMENTAL — Lung recruitment maneuver (LRM) is a transitory and controlled increase in airway pressure to open collapsed alveoli. LRM is the first step of the PEEP DECREMENTAL method. After LRM, PEEP is systematically decreased, in small decrements, until the best respiratory system mechanics is identified.
  Other Names: PEEP_Titration

SUMMARY:
The goal of this interventional crossover study in morbidly obese intubated and mechanically ventilated patients is to describe the respiratory mechanics and the heart-lung interaction at titrated positive end-expiratory pressure levels following a recruitment maneuver with transthoracic echocardiography and electric impedance tomography imaging.

DETAILED DESCRIPTION:
Obese patients under mechanical ventilation are more likely to develop atelectasis as a consequence of the increased abdominal weight. Atelectasis is the primary responsible for respiratory insufficiency and impossibility to wean obese patients from respiratory support.

In a previous study we demonstrated the efficacy of the application of titrated PEEP levels following a recruitment maneuver in obese patients, i.e. improvement in respiratory mechanics and gas exchanges without negative hemodynamic effects.

The application of lung and heat imaging will allow us to quantitatively describe:

* Increase in aerated lung tissue (reduction of atelectasis)
* Reduction of over-inflation of the ventilated regions
* Recoupling of ventilation and perfusion
* Improvement in right heart function by reduction of right heart afterload

ELIGIBILITY:
Inclusion Criteria:

* ICU admitted requiring intubation and mechanical ventilation
* BMI ≥ 35 kg/m2
* Waist circumference > 88 cm (for women)
* Waist circumference > 102 cm (for men)

Exclusion Criteria:

* Known presence of esophageal varices
* Recent esophageal trauma or surgery
* Severe thrombocytopenia (Platelets count ≤ 5,000/mm3)
* Severe coagulopathy (INR ≥ 4)
* Presence or history of pneumothorax
* Pregnancy
* Patients with poor oxygenation index (PaO2/FiO2< 100 mmHg with at least 10 cmH2O of PEEP)
* Pacemaker and/or internal cardiac defibrillator
* Hemodynamic parameters: systolic blood pressure (SBP) <100 mmHg and >180 mmHg, or if SBP is between 100-180 mmHg on high dose of IV continuous infusion norepinephrine (>20 μg per minute), or dobutamine (>10 μg per minute), or dopamine (>10 μg per Kg per minute), or epinephrine (>10 μg per minute).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-04; Primary Completion 2021-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Respiratory System Elastance | During study time points :baseline, PEEP incremental, PEEP decremental
  Difference in Respiratory System Elastance measured in cmH2O/L

SECONDARY OUTCOMES:
Lung mechanics - Compliance | Study time points: baseline, PEEP incremental, PEEP decremental
  Difference in respiratory system, lung and chest wall compliance measured in mL/cmH2O
Lung mechanics - Airway resistances | During study time points: baseline, PEEP incremental, PEEP decremental
  Difference in resistances of the airways measured as cmH2O/L/sec (Raw)
Survival | 28 days after the performance of the study protocol
  Incidence of death among the study population

OTHER OUTCOMES:
Intra-abdominal pressure | Study time point: baseline
  Changes in bladder pressure measured in mmHg.
Electrical Impedance Tomography measurement: collapsed and overdistension | Study time points: baseline, PEEP incremental, PEEP decremental
  Percentage of lung tissue collapsed and over distended at different PEEP levels by analyzing pixel compliance ( variation in impedance divided by applied pressure during a respiratory cycle).
Electrical Impedance Tomography measurement: distribution of ventilation | Study time points: baseline, PEEP incremental, PEEP decremental
  Difference in end-expiratory lung impedance as percentage estimating the distribution of ventilation among 4 horizontal regions of interest ( from non-dependent to dependent lung regions).
Electrical Impedance Tomography measurement: lung perfusion | Study time points: baseline, PEEP incremental, PEEP decremental
  Differences in distribution in lung perfusion measured as regional percentage of the total cardiac output.
Central venous pressure | Study time points: baseline, PEEP incremental, PEEP decremental. Follow up: 1, 2 , 24 and 48 hours after study procedures
  Changes in central venous pressure (CVP, mmHg)
Gas Exchange - Oxygenation | Study time points: baseline, PEEP incremental, PEEP decremental. Follow up: 1, 2 , 24 and 48 hours after study procedures
  Difference in oxygenation measured in mmHg of PaO2/FiO2
Gas Exchange - Arterial carbon dioxide | Study time points: baseline, PEEP incremental, PEEP decremental. Follow up: 1, 2 , 24 and 48 hours after study procedures
  Difference in arterial carbon dioxide measured in mmHg (PaCO2)
Lung volumes - respiratory dead space | Study time points: baseline, PEEP incremental, PEEP decremental.
  Difference in dead space fraction measured as the ratio of death volume over the total tidal volume (Vd/Vt)
Heart rate | Study time points: baseline, PEEP incremental, PEEP decremental. Follow up: 1, 2 , 24 and 48 hours after study procedures
  Changes in heart rate (HR, bpm)
Blood pressure | A) 48 and 24h before study procedures B)Study time points: baseline, PEEP incremental, PEEP decremental C)Follow up: 1, 2 , 24, 48 and 72 hours after study procedures.
  Changes in invasive arterial blood pressures (BP, mmHg)
Right heart function -Tricuspid Annular Plane Systolic Excursion (TAPSE) | Study time points: baseline, PEEP incremental, PEEP decremental. Follow up: 1, 2 , 24 and 48 hours after study procedures
  Differences in TAPSE measured through two-dimensional transthoracic echocardiography (apical four-chamber view).
Right heart function - S' | Study time points: baseline, PEEP incremental, PEEP decremental. Follow up: 1, 2 , 24 and 48 hours after study procedures
  Differences in the systolic excursion of the tricuspid annulus measured by tissue doppler imaging.
Right heart function - Tei index | Study time points: baseline, PEEP incremental, PEEP decremental
  Differences in global right ventricular function obtained from right ventricle tissue doppler imaging.
Vasopressor requirement | 48, 24h before AND 24, 48 and 72h after study procedures.
  Norepinephrine (mcg/kg/min), epinephrine (mcg/kg/min) , phenylephrine ( mcg/kg/min) and vasopressin (U / min)
Creatinine | 48, 24h before AND 24, 48 and 72h after study procedures.
  Serum level of creatinine
Urinary output | 48, 24h before AND 24, 48 and 72h after study procedures.
  Changes in urinary output (mL)
Fluid balance | 48, 24h before AND 24, 48 and 72h after study procedures.
  Changes in fluid balance (mL)
Incidence of tracheostomy | 28 days after the performance of the study protocol
  Necessity of tracheostomy for prolonged ventilatory support among the study population
Duration of mechanical ventilation | 28 days after the performance of the study protocol
  Number of days on mechanical ventilation
Intensive care unit length of stay | 28 days after the performance of the study protocol
  Numbers of days spent in the intensive care
Hospital length of stay | 28 days after the performance of the study protocol
  Numbers of days spent in the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kacmarek, RRT, PhD, Principal Investigator — Massachusetts General Hospital; Lorenzo Berra, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Akoumianaki E, Maggiore SM, Valenza F, Bellani G, Jubran A, Loring SH, Pelosi P, Talmor D, Grasso S, Chiumello D, Guerin C, Patroniti N, Ranieri VM, Gattinoni L, Nava S, Terragni PP, Pesenti A, Tobin M, Mancebo J, Brochard L; PLUG Working Group (Acute Respiratory Failure Section of the European Society of Intensive Care Medicine). The application of esophageal pressure measurement in patients with respiratory failure. Am J Respir Crit Care Med. 2014 Mar 1;189(5):520-31. doi: 10.1164/rccm.201312-2193CI. PMID 24467647
- [Background] Behazin N, Jones SB, Cohen RI, Loring SH. Respiratory restriction and elevated pleural and esophageal pressures in morbid obesity. J Appl Physiol (1985). 2010 Jan;108(1):212-8. doi: 10.1152/japplphysiol.91356.2008. Epub 2009 Nov 12. PMID 19910329
- [Background] Borges JB, Suarez-Sipmann F, Bohm SH, Tusman G, Melo A, Maripuu E, Sandstrom M, Park M, Costa EL, Hedenstierna G, Amato M. Regional lung perfusion estimated by electrical impedance tomography in a piglet model of lung collapse. J Appl Physiol (1985). 2012 Jan;112(1):225-36. doi: 10.1152/japplphysiol.01090.2010. Epub 2011 Sep 29. PMID 21960654
- [Background] Reinius H, Jonsson L, Gustafsson S, Sundbom M, Duvernoy O, Pelosi P, Hedenstierna G, Freden F. Prevention of atelectasis in morbidly obese patients during general anesthesia and paralysis: a computerized tomography study. Anesthesiology. 2009 Nov;111(5):979-87. doi: 10.1097/ALN.0b013e3181b87edb. PMID 19809292
- [Background] Victorino JA, Borges JB, Okamoto VN, Matos GF, Tucci MR, Caramez MP, Tanaka H, Sipmann FS, Santos DC, Barbas CS, Carvalho CR, Amato MB. Imbalances in regional lung ventilation: a validation study on electrical impedance tomography. Am J Respir Crit Care Med. 2004 Apr 1;169(7):791-800. doi: 10.1164/rccm.200301-133OC. Epub 2003 Dec 23. PMID 14693669
- [Background] Costa EL, Lima RG, Amato MB. Electrical impedance tomography. Curr Opin Crit Care. 2009 Feb;15(1):18-24. doi: 10.1097/mcc.0b013e3283220e8c. PMID 19186406
- [Background] Krishnan S, Schmidt GA. Acute right ventricular dysfunction: real-time management with echocardiography. Chest. 2015 Mar;147(3):835-846. doi: 10.1378/chest.14-1335. PMID 25732449
- [Background] Vieillard-Baron A, Jardin F. Why protect the right ventricle in patients with acute respiratory distress syndrome? Curr Opin Crit Care. 2003 Feb;9(1):15-21. doi: 10.1097/00075198-200302000-00004. PMID 12548024
- [Derived] De Santis Santiago R, Teggia Droghi M, Fumagalli J, Marrazzo F, Florio G, Grassi LG, Gomes S, Morais CCA, Ramos OPS, Bottiroli M, Pinciroli R, Imber DA, Bagchi A, Shelton K, Sonny A, Bittner EA, Amato MBP, Kacmarek RM, Berra L; Lung Rescue Team Investigators. High Pleural Pressure Prevents Alveolar Overdistension and Hemodynamic Collapse in Acute Respiratory Distress Syndrome with Class III Obesity. A Clinical Trial. Am J Respir Crit Care Med. 2021 Mar 1;203(5):575-584. doi: 10.1164/rccm.201909-1687OC. PMID 32876469